CLINICAL TRIAL: NCT02835274
Title: Directional Lead: Investigation of Rotational Current Steering, Ease of Use of Clinical Effects Map, and Therapeutic Outcomes of Deep Brain Stimulation
Brief Title: Study to Characterize Acute and Chronic Directional Aspects of Deep Brain Stimulation
Acronym: DIRECT-DBS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: A4150
Record Dates: First submitted 2016-06-24; First posted 2016-07-18 (Estimated); Results first posted 2020-02-07 (Actual); Last update posted 2020-11-19 (Actual); Status verified 2020-11

CONDITIONS: Parkinson Disease
Keywords: parkinson disease; deep brain stimulation; directional stimulation
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ring mode followed by Unrestricted mode (Experimental): omni-directional stimulation followed by unrestricted Mode stimulation
  Interventions: Device: BSC Deep Brain Stimulation System with Directional Lead
- Unrestricted mode followed by ring mode (Active Comparator): Unrestricted Mode stimulation followed by omni-directional stimulation
  Interventions: Device: BSC Deep Brain Stimulation System with Directional Lead

INTERVENTIONS:
Device: BSC Deep Brain Stimulation System with Directional Lead

SUMMARY:
The primary objective is to characterize the programming effects of Boston Scientific Vercise™ PC System using the DBS Directional Lead for bilateral STN DBS for the treatment of Parkinson's disease in acute and chronic settings.

ELIGIBILITY:
Key Inclusion Criteria:

* Diagnosis of bilateral idiopathic PD with the presence of rigidity and at least one (1) of the following: resting tremor or bradykinesia.
* UPDRS III score of >25 in the meds OFF condition
* Medication must improve PD symptoms by ≥30%, as measured by UPDRS subset III score

Key Exclusion Criteria:

* Any significant psychiatric problems, including unrelated clinically significant depression as determined by the investigator
* Any current drug or alcohol abuse as determined by the investigator
* Any history of recurrent or unprovoked seizures
* Any significant medical condition that is likely to interfere with study procedures or likely to confound evaluation of study endpoints, including any terminal illness with survival <12 months

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2016-07-19 (Actual); Primary Completion 2018-12-19 (Actual); Study Completion 2018-12-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roshini Jain, Study Director — Boston Scientific Neuromodulation Corporation
Locations (3):
- CHU Grenoble - Hopital Michallon, Grenoble, France
- Universitaetsklinikum Wuerzburg, Würzburg, Germany
- Academisch Medisch Centrum, Amsterdam, Netherlands

RESULTS

PARTICIPANT FLOW:
Groups:
- Ring Mode Followed by Unrestricted Mode: omni-directional stimulation followed by unrestricted Mode stimulation
  BSC Deep Brain Stimulation System with Directional Lead
- Unrestricted Mode Followed by Ring Mode: Unrestricted Mode stimulation followed by omni-directional stimulation
  BSC Deep Brain Stimulation System with Directional Lead
Period: Overall Study
Arm/Group | Ring Mode Followed by Unrestricted Mode | Unrestricted Mode Followed by Ring Mode
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ring Mode Followed by Unrestricted Mode | Unrestricted Mode Followed by Ring Mode | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 66 (9) | 61 (6) | 63.4 (7.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 4
  Male | 5 | 3 | 8
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Unified Parkinson's Disease Rating Scale (UPDRS) Scores - Motor Section (Part III) at End of Randomized Phase
Description: Mean change in Unified Parkinson's Disease Rating Scale (UPDRS) scores - motor section (Part III) at end of randomized phase in meds ON condition
  Range of UPDRS III is 0 - 108 with greater scores indicating worse disease state
Time Frame: Up to 12 months post-implant
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Ring Mode; Unrestricted Mode: BSC Deep Brain Stimulation System with Directional Lead
Arm/Group | Ring Mode | Unrestricted Mode
Number analyzed (Participants) | 12 | 12
units on a scale
  Baseline | 21 (11) | 21 (11)
  End of Randomized Phase | 13 (8) | 16 (10)

ADVERSE EVENTS:
Time Frame: Adverse events up to end of randomized phase (~ up to 120 days post implant)
Description: Adverse events up to end of randomized phase
Groups:
- Ring Mode: Ring Mode
  BSC Deep Brain Stimulation System with Directional Lead
- Unrestricted Mode: Unrestricted mode
  BSC Deep Brain Stimulation System with Directional Lead
Arm/Group | Ring Mode | Unrestricted Mode
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-02-25): https://cdn.clinicaltrials.gov/large-docs/74/NCT02835274/Prot_SAP_000.pdf